CLINICAL TRIAL: NCT06029842
Title: A Randomized Controlled Trial to Assess the Role of a Clinical Pharmacist in the Management of Type 2 Diabetic Patients for Optimum Treatment Outcomes in a Primary Medical Center in Jordan
Brief Title: The Role of a Clinical Pharmacist in the Management of Type 2 Diabetic Patients in a Primary Medical Center in Jordan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Jyana Alelaimat, Master student at the University of Jordan, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Clinical pharmacist
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-10

CONDITIONS: Pharmacist-Patient Relations
Keywords: clinical pharmacist; medical center; Ministry of Health; Collaborative approach
MeSH Terms: interventions — Physicians

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- the intervention group (Other): this group received the collaborative care between the clinical pharmacist and physicians in a medical center
  Interventions: Other: Collaborative approach of clinical pharmacist with physicians in a medical center
- the control group (No Intervention): this group received the standard care of physicians in a medical center without clinical pharmacist interventions

INTERVENTIONS:
Other: Collaborative approach of clinical pharmacist with physicians in a medical center — For those who allocated to the intervention group, the clinical pharmacist interviewed them at each monthly visit about 30 minutes before seeing physicians, the clinical pharmacist identified treatment related problems, provided medication counseling, answered questions asked by patients or physicians, encouraged compliance, offered instructions on self-monitoring of blood pressure and glucose levels, distributed educational materials about diabetes and emphasis was made on optimizing adherence to pharmacological and non- pharmacological therapy. the pharmacist interventions on treatment related problems (TRPs) and proposed patient care plans were discussed with treatng physicians who decided to accept or reject them.
  Arms: the intervention group

SUMMARY:
This study aimed to assess the impact of the clinical pharmacist on enhancing type 2 diabetic patients outcomes in a primary health care center.

DETAILED DESCRIPTION:
About 103 patients with type 2 diabetes were randomized to control or intervention group, the control group received a standard care, while the intervention group received the collaborative care between the clinical pharmacist and physicians. Fasting blood glucose, HbA1c, Lipid profile, and blood pressure measured for both groups at baseline and after three months of follow-up. Treatment related problems (TRPs), quality of life, adherence, and patients knowledge about their medications were assessed. Cost avoidance and clinical significance of implemented clinical pharmacist interventions were assessed too.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetic patients who aged 18 years or more with a HbA1c reading 6.5 % or more at the time of diagnosis

Exclusion Criteria:

* pregnant patients
* breastfeeding patients
* patients with urgent or emergent cases
* patients with cognitive impairment
* if the patient is unable to provide informed written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-04-24 (Actual)

PRIMARY OUTCOMES:
HbA1c | 3 months

SECONDARY OUTCOMES:
Lipid profile | 3 months
  LDL , HDL , TGS
Fasting blood glucose | each month for 3 months
Patients knowledge about their medications | 3 months
  Validated questionnaire were used. According to Abu Farha et.al, Patients' medication knowledge was assessed by their ability to answer correctly the questions related to their medication doses, indications and timing. For each correct statement the patient gained 1 point with a total of 3 points for each medication. Patients were considered to have suboptimal knowledge if they obtain an average medication score of 2 or less.
Cost avoidance of implemented clinical pharmacist interventions | 3 months
  The cost avoidance of implemented interventions were evaluated relevant to "presumed cost avoidance". This implies an action that reduces or eliminates additional spending that would have happened if the intervention had not occurred. The reduction in costs was estimated using the cost avoidance values that were derived from Campbell. The resulting cost avoidance values for individual clinical pharmacy intervention types are listed below for individual clinical pharmacy intervention type.* Intervention type, Overall cost avoidance, $ Addition of a medication 62.81
  * Change medication 74.67
  * Discontinuation of a medication 57.25
  * Dosage form change 67.33
  * Dose adjustment 71.41
  * Drug information 26.97
  * Medication reconciliation 472.86
  * Monitoring laboratory order 93.58
  * Non-formulary consultation 56
  * Non-formulary to formulary conversion 44
  * Pharmacokinetic monitoring-level adjustment 91.08
  * Prevention of adverse drug event 581.08
  * Prompted medical follow-up 70.33
Patients adherence to medications | 3 months
  Patients' adherence to medications was assessed by Oriana Awwad et al.2022 validated Arabic version of the Morisky, Green, and Levine (MGL) adherence scale [16], This scale is "a 4-item instrument used to identify patients with chronic disease who are not taking their medications as prescribed". The scale encloses four questions: 1) "Do you ever forget to take your medicine?" 2) "Are you careless at times about taking your medicine?" 3) "When you feel better do you sometimes stop taking your medicine?" and 4) "Sometimes if you feel worse when you take the medicine, do you stop taking it?" It has a scoring scheme of "Yes" = 1 and "No" = 0 for each item with a total score ranging from 0 to 4. The sum of "Yes" answers provides a composite measure of non-adherence. Lower evaluations imply a higher level of adherence, and total patient scores can be classified into high adherence level (0 answered "yes"), moderate adherence level (1-2 answered "yes") and low level adherence (3-4 "yes").
Quality of life | 3 months
  The change in the Quality of Life questionnaire (EQ-5D-5L) was assessed. At baseline, all patients were asked to self-complete the Quality of Life (EQ-5D-5L) questionnaire. This self-completed questionnaire consists of 5 domains" (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression)" in which each dimension is rated with 5 levels of severity (no problems, slight problems, moderate problems, severe problems, and unable to perform or extreme problems). The answers on these domains are translated to give a consequent number; e.g 23445. These numbers have a health utility index score which already had been studied and validated for different population in a number of countries. A single index value for all health states with a range from 0 (where zero is a health state equivalent to death). Another factor express QoL is EQ-vas which is a scale from 0 to 100 where the patients are asked to indicate their overall health on the day after completion of questionnair.
Blood pressure | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Abu-Nsair medical center, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Yes